CLINICAL TRIAL: NCT06679491
Title: Effects of Menstrual Cycle-based Undulating Periodized Resistance Training in Women's Neuromuscular Abilities
Brief Title: Impact of Menstrual Cycle-Based Resistance Training on Neuromuscular Performance in Female Athletes
Acronym: MENSES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universite de La Reunion (Other)
Collaborators: Physio Formation (Unknown)
Responsible Party: Principal Investigator, Manon DAUVERGNE, PhD Candidate, Universite de La Reunion
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ULaReunion; AU1941 - 24.00913.000257 (Other: Comité de Protection des Personnes Sud-est IV)
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Menstrual Cycle; Resistance Training; Neuromuscular Function; Female Athlete; Women Health; Oral Contraceptive Pill; Muscle Strenght; Hormones; Periodized Training
Keywords: Menstrual Cycle; Resistance training; Periodized training; neuromuscular function; Female athlete; Hormones; oral contraceptive pill; women health

STUDY DESIGN:
Intervention Model Description: This study uses a parallel-group, randomized, controlled interventional model with four arms. Participants are allocated to one of four groups based on menstrual cycle status and training intensity patterns:
  Three groups consist of female athletes with natural menstrual cycles who are assigned to different training regimens based on specific menstrual phases (higher intensity in either follicular or luteal phases, or a continuous approach).
  The fourth group includes female athletes on oral contraceptives who follow a continuous training regimen as a control.
  Each participant completes a 13-week resistance training program with two weekly sessions. Randomization is stratified by BMI and age to ensure balanced group characteristics. The primary objective is to assess changes in neuromuscular function, with each group experiencing variations in training intensity aligned with hormonal influences across menstrual phases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- N-PF (Natural Cycle - Follicular Phase-Intensified Training) (Experimental): Female athletes with natural menstrual cycles who follow a resistance training program with increased intensity during the follicular phase and reduced intensity during the luteal phase. This arm aims to evaluate the impact of follicular-phase-focused training on neuromuscular performance, leveraging the potential effects of elevated estrogen levels during this phase.
  Intervention:
  Resistance Training Program: 13 weeks, 2 sessions per week, with higher intensity training scheduled during the follicular phase (early and late) and reduced intensity during the luteal phase.
  Interventions: Other: Resistance periodized training program (N-PF)
- N-PL (Natural Cycle - Luteal Phase-Intensified Training) (Experimental): Description: Female athletes with natural menstrual cycles who undergo a resistance training program with increased intensity during the luteal phase and reduced intensity during the follicular phase. This approach assesses the impact of training when progesterone levels are elevated.
  Intervention:
  Resistance Training Program: 13 weeks, 2 sessions per week, with higher intensity training during the luteal phase (early and late) and reduced intensity during the follicular phase.
  Interventions: Other: Resistance peioridized training program (N-PL)
- N-C (Natural Cycle - Continuous Training) (Experimental): Description: Female athletes with natural menstrual cycles who participate in a continuous intensity training program across all phases of the menstrual cycle. This group provides a comparison to determine the effects of a non-phase-specific training protocol on neuromuscular function.
  Intervention:
  Resistance Training Program: 13 weeks, 2 sessions per week, maintaining a consistent training intensity across both follicular and luteal phases.
  Interventions: Other: Continuous resistance training program (C)
- OCP-C (Oral Contraceptive - Continuous Training, Control Group) (Active Comparator): Description: Female athletes using oral contraceptives, following a continuous intensity training program regardless of menstrual phase. This group serves as a control, providing insight into the neuromuscular effects of training under the hormonal conditions set by oral contraceptive use.
  Intervention:
  Resistance Training Program: 13 weeks, 2 sessions per week, with continuous intensity across all training sessions due to the stable hormonal environment induced by oral contraceptives.
  Interventions: Other: Continuous resistance training program (C)

INTERVENTIONS:
Other: Resistance periodized training program (N-PF) — This intervention consists of a 13-week structured resistance training program tailored to align with the natural menstrual cycle, focusing on intensified training during the follicular phase. Participants perform two resistance training sessions per week, each lasting 90 minutes, with intensity modulated based on the participant's menstrual phase.
  Intensity Modulation:
  Follicular Phase (Days 1-14): Training sessions are performed at a higher training load during both early and late follicular phases. The increased intensity leverages higher estrogen levels, which may support greater muscle strength and recovery during this phase.
  Luteal Phase (Days 15-28): Training sessions are conducted at a lower training load during both early and late luteal phases to accommodate the hormonal shifts associated with elevated progesterone.
  Arms: N-PF (Natural Cycle - Follicular Phase-Intensified Training)
Other: Resistance peioridized training program (N-PL) — This intervention consists of a 13-week structured resistance training program tailored to align with the natural menstrual cycle, focusing on intensified training during the luteal phase. Participants perform two resistance training sessions per week, each lasting 90 minutes, with intensity modulated according to the participant's menstrual phase.
  Intensity Modulation:
  Follicular Phase (Days 1-14): Training sessions are conducted at a lower training load during both early and late follicular phases to accommodate the hormonal environment of this phase.
  Luteal Phase (Days 15-28): Training sessions are performed at a higher training load during both early and late luteal phases. The increased intensity leverages the hormonal environment associated with elevated progesterone, which may affect muscle endurance and neuromuscular adaptations during this phase.
  Arms: N-PL (Natural Cycle - Luteal Phase-Intensified Training)
Other: Continuous resistance training program (C) — This intervention consists of a 13-week structured resistance training program with a continuous training intensity maintained throughout the menstrual cycle. Participants perform two resistance training sessions per week, each lasting 90 minutes, with a consistent training load applied across all phases.
  Intensity Modulation:
  All Phases: Training sessions are conducted at a steady training load regardless of menstrual phase. This continuous approach is designed to provide a baseline for assessing neuromuscular adaptations without the influence of phase-specific intensity adjustments.
  Arms: N-C (Natural Cycle - Continuous Training); OCP-C (Oral Contraceptive - Continuous Training, Control Group)

SUMMARY:
The goal of this clinical trial is to assess the impact of menstrual cycle-based resistance training on neuromuscular function in female athletes.

The primary questions it aims to answer are :

* Does varying resistance training intensity according to menstrual phases improve maximal knee extensor strength?
* How do different training protocols affect voluntary activation, rate of force development, muscle stiffness, and vertical jump height?

Researchers will compare natural menstrual cycle groups with an oral contraceptive control group to determine if menstrual phase-specific training influences neuromuscular adaptations.

Participants will:

* Undergo 2 weekly resistance training sessions over 13 weeks with intensity adjustments based on menstrual phase
* Complete periodic neuromuscular assessments across three menstrual phases: early follicular, late follicular, and mid-luteal before and after resistance training intervention

DETAILED DESCRIPTION:
This study investigates the neuromuscular effects of menstrual cycle-based resistance training by comparing three distinct training protocols among female athletes with natural menstrual cycles and a control group of athletes using oral contraceptives. Hormonal fluctuations across the menstrual phases can impact muscle performance, recovery, and neuromuscular function. This trial aims to align training intensity with menstrual cycle phases to enhance neuromuscular adaptations.

Study Design and Population

The trial is a controlled, randomized, open-label design involving 60 recreationally active female athletes aged 18 and above. Participants are allocated into four groups:

N-PF: Natural menstrual cycle with increased training intensity during the follicular phase.

N-PL: Natural menstrual cycle with increased training intensity during the luteal phase.

N-C: Natural menstrual cycle with continuous training intensity across all phases.

OCP-C: Oral contraceptive users with continuous training intensity. Each participant completes a 13-week resistance training program tailored to her group's specific phase-aligned training protocol, with two sessions per week. To assess the neuromuscular impact, we perform pre- and post-intervention evaluations across three key menstrual phases: early follicular, late follicular, and mid-luteal.

Neuromuscular Assessments Primary outcomes include maximal knee extensor strength, assessed through isokinetic testing, and secondary measures cover neuromuscular activation, rate of force development (RFD), muscle stiffness, and vertical jump performance (CMJ). These assessments are conducted during each of the three menstrual phases pre- and post-intervention to capture phase-specific neuromuscular adaptations. Blood sampling for hormonal verification (estradiol and progesterone levels) accompanies each phase-specific testing session.

Methodology and Rationale The training intensity and volume are adjusted based on the participant's menstrual phase to leverage hormonal benefits, with estrogen levels typically promoting muscular strength in the follicular phase and progesterone affecting endurance in the luteal phase. We hypothesize that phase-specific training may yield greater improvements in strength, muscle stiffness, and overall neuromuscular efficiency.

This study's findings are expected to provide novel insights into optimizing training loads for female athletes according to hormonal cycles, with implications for improving performance, reducing injury risk, and advancing individualized training and rehabilitation protocols.

ELIGIBILITY:
Inclusion Criteria:

* Female athletes with natural menstrual cycles (eumenorrheic): Participants must have regular menstrual cycles lasting between 21 and 35 days, with at least 9 cycles per year.
* Women using a low-dose monophasic estrogen-progestin oral contraceptive.
* Age 18 or older: Participants must be legal adults.
* Body Mass Index (BMI) between 18 and 30 kg/m².
* No medical contraindications to high-level physical training or exercise.
* Physically active: Engages in at least 3 hours of physical activity per week.
* Informed consent: Provides written, informed consent to participate in the study.
* Affiliation with a social security system (if applicable by local regulations).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal knee extensor strenght | From baseline assessment prior to intervention to post-intervention at 13 weeks.
  Description:
  This outcome measure assesses the maximal isokinetic strength of the knee extensor muscles, measured as peak torque (rotational force) in Newton-meters (Nm), using an isokinetic dynamometer.
  Scoring and Interpretation:
  Higher scores indicate greater strength, with no theoretical upper limit as scores are determined by the individual's maximal voluntary contraction.
  Typical Range: In athletic populations, peak torque values generally range from 100 to 250 Nm, but individual results may vary based on factors like muscle size and training status.
  Criteria for Change: An improvement in peak torque post-intervention indicates a positive neuromuscular adaptation to the training program.
  This measure quantifies changes in lower limb strength over time, allowing comparison of neuromuscular adaptations between menstrual phase-aligned and continuous training groups.

SECONDARY OUTCOMES:
Rate of Force Development (RFD) | From baseline assessment prior to intervention to post-intervention at 13 weeks
  Evaluates the speed at which force is generated by the knee extensor muscles. This is a key indicator of explosive strength, relevant for sports performance.
  Measurement: Calculated as the slope of the force-time curve from the onset of muscle contraction.
  Relevance: Higher RFD values suggest improved neuromuscular response and power output.
Active muscle stiffness | From baseline assessment prior to intervention to post-intervention at 13 weeks.
  Measures the active stiffness of the knee extensor muscles during before and after a fatiguing task, at 50%MVC with a shear wave elastrography (SWE) methods.
Voluntary Muscle Activation (%AV) | From baseline assessment prior to intervention to post-intervention at 13 weeks.
  Description: Assesses the degree of maximal voluntary activation in the knee extensor muscles before, during and after an "all-out" effort. This test captures the participant's capacity to recruit motor units fully, measured using twitch interpolation technique to evaluate the difference between voluntary and stimulated muscle force output.
  Relevance: This measure reflects the participant's neuromuscular efficiency by indicating their ability to achieve maximal muscle activation without additional external stimulation. It provides insight into central nervous system drive and the efficiency of motor unit recruitment during intense exertion.
Vertical Jump Height (Countermovement Jump - CMJ) | From baseline assessment prior to intervention to post-intervention at 13 weeks.
  Measures the maximal height achieved during a countermovement jump, recorded as a functional measure of lower body power. Relevance: Vertical jump height reflects overall lower limb strength and power, providing insight into functional athletic performance.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas PEYROT, Professor (PU), Study Director — Université du Mans; Manon DAUVERGNE, Professor (Assistant), Study Director — Universite de La Reunion
Locations (1):
- Laboratoire IRISSE (Université de La Réunion), Le Tampon, France, Reunion

IPD SHARING:
Plan to Share IPD: Undecided